CLINICAL TRIAL: NCT00278902
Title: A Study of ARRY-334543 in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Array Biopharma, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Array BioPharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARRY-0501
Record Dates: First submitted 2006-01-17; First posted 2006-01-19 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Advanced Cancer
Keywords: ErbB2+ Breast Cancer; HER2+ Breast Cancer
MeSH Terms: interventions — ARRY-334543

ARMS (1):
- ARRY-334543 (Experimental)
  Interventions: Drug: ARRY-334543, EGFR/ErbB2 inhibitor; oral

INTERVENTIONS:
Drug: ARRY-334543, EGFR/ErbB2 inhibitor; oral — Part 1: single dose and multiple dose, escalating; Part 2: multiple dose, single schedule

SUMMARY:
This is a Phase 1 study during which patients with advanced solid tumors will receive investigational study drug ARRY-334543.

This study has 2 parts. In the first part, patients will receive increasing doses of study drug (2 dosing schedules will be evaluated) in order to achieve the highest dose possible that will not cause unacceptable side effects. Approximately 70 patients from the US and Canada will be enrolled in Part 1 (Completed).

In the second part of the study, patients will receive the best dose(s) and schedule(s) of study drug determined from the first part of the study and will be followed to see what side effects the study drug causes and what effectiveness it has, if any, in treating the cancer. Approximately 40 patients from the US and Canada will be enrolled in Part 2 (Completed).

ELIGIBILITY:
Key Inclusion Criteria (Part 2):

* Histologically or cytologically confirmed diagnosis of ErbB2+ breast cancer, pancreatic, squamous cell head and neck, hepatocellular, hepatobiliary, glioblastoma, ovarian, prostate, upper GI, colorectal, non small cell lung, or bladder cancer or other relevant cancers if approved in advance by the Sponsor.
* Measurable disease (at least 1 target lesion) according to modified RECIST.
* Failed at least one previous therapeutic regimen and either no longer a candidate for standard therapy, has no standard therapy available, or chooses not to pursue standard therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.
* Must consent to allow the Sponsor access to an archival histological specimen or to have a pre-dose tumor biopsy.
* Additional criteria exist.

Key Exclusion Criteria (Part 2):

* Uncontrolled or symptomatic brain metastases (if a patient has brain metastases and is on steroids, the steroid dose must be stable for at least 30 days).
* Use of an investigational medication or device within 30 days prior to first dose of study drug.
* Major surgery within 30 days prior to first dose of study drug.
* Radiotherapy or chemotherapy within 28 days prior to first dose of study drug (not including palliative radiotherapy at focal sites).
* Pregnancy or lactation.
* Known positive serology for the human immunodeficiency virus (HIV), hepatitis B and/or hepatitis C. Of note, if a patient has hepatocellular carcinoma, then they may be enrolled even if they are positive for hepatitis B and/or hepatitis C.
* Additional criteria exist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2006-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Establish the maximum tolerated dose (MTD) of study drug. | Part 1
Characterize the safety profile of the study drug in terms of adverse events, clinical laboratory tests, vital signs and electrocardiograms. | Part 1 and Part 2

SECONDARY OUTCOMES:
Characterize the pharmacokinetics (PK) of the study drug in terms of plasma concentrations. | Part 1 and Part 2
Assess the efficacy of the study drug in terms of tumor dimension assessment. | Part 1 and Part 2

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- United States (3):
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon Research Center, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Canada (2):
  - British Columbia Cancer Agency- Centre for the Southern Interior, Kelowna, British Columbia
  - British Columbia Cancer Agency, Vancouver, British Columbia